CLINICAL TRIAL: NCT03760874
Title: Prospective Register Study to Record Safety and Efficacy of Oral Anticoagulants in Atrial Fibrillation Patients
Brief Title: Atrial Fibrillation Research Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, MD, PhD, Assistant Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 19062013
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anticoagulants and Bleeding Disorders; Atrial Fibrillation
MeSH Terms: conditions — Hemostatic Disorders; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non Vitamin K Oral Anticoagulant: Dabigatran, Rivaroxaban, Apixaban, Edoxaban
- Vitamin K Oral Anticoagulant: Warfarin, Acenocoumarol.

SUMMARY:
All patients with atrial fibrillation who are treated with vitamin-k antagonists (warfarin, phenprocoumon) or non vitamin K oral anticoagulants (Dabigatran, Rivaroxaban, Apixaban, Edoxaban) in real world settings will be recorded in this register. Within this register a characterization of patients and therapy (with regard to medication, dose and duration) will be done. On basis of defined clinical relevant end points the long-term efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation
* Indication for oral anticoagulant treatment

Exclusion Criteria:

* Missing Informed Consent Form
* Missing Contact Informations for Follow up

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with atrial fibrillation in clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-06-13 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic Events | 1 year
Bleeding Events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russo V, Carbone A, Attena E, Rago A, Mazzone C, Proietti R, Parisi V, Scotti A, Nigro G, Golino P, D'Onofrio A. Clinical Benefit of Direct Oral Anticoagulants Versus Vitamin K Antagonists in Patients with Atrial Fibrillation and Bioprosthetic Heart Valves. Clin Ther. 2019 Dec;41(12):2549-2557. doi: 10.1016/j.clinthera.2019.10.008. Epub 2019 Nov 14. PMID 31735436